CLINICAL TRIAL: NCT05776381
Title: The Impact of an In-consultation Patient Decision Aid on Treatment Choices and Outcomes of Management for Patients With an Unexpected Malignant Colorectal Polyp A Non-randomized Clinical Phase II Study
Brief Title: The Impact of a Patient Decision Aid on Treatment Choices for Patients With an Unexpected Malignant Colorectal Polyp
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SDM in malignant polyps
Record Dates: First submitted 2023-03-02; First posted 2023-03-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Shared Decision Making; Colonic Polyp; Decision Aids; Rectal Polyp; Colorectal Polyp; Colorectal Cancer
Keywords: non-randomized trial; malignant colorectal polyp; Patient Decision aid; Shared Decision Making
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a clinical multicenter, non-randomized, interventional phase II study. Three to five departments of colorectal surgery in Danish hospitals will be invited to participate in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making (SDM) (Experimental): Patients with an unexpected malignant colorectal polyp where a decision needs to be made concerning the management of care.
  Interventions: Other: Shared Decision Making using a Patient Decision Aid.
- Historical data arm (No Intervention): Historical data on the management of patients with an unexpected malignant colorectal polyp from February 2018 to the end of 2022 retrieved through the Danish Colorectal Cancer Group Database, the National Pathology database and the National Patient Register.

INTERVENTIONS:
Other: Shared Decision Making using a Patient Decision Aid. — The intervention comprises the surgeon actively using the tailored PtDA and SDM with the patient when deciding on the management of an unexpected malignant colorectal polyp.
  Arms: Shared Decision Making (SDM)

SUMMARY:
Management of unexpected malignant colorectal polyps removed endoscopically can be challenging due to the risk of residual tumor and lymphatic spread. International studies have shown that in patients choosing surgical management instead of watchful waiting, 54-82% of bowel resections are without evidence of residual tumor or lymphatic spread. As surgical management entails risks of complications and watchful waiting management entails risks of residual disease or recurrence, a clinical dilemma arises when choosing a management strategy.

Shared decision making (SDM) is a concept that can be used in preference sensitive decision making to facilitate patient involvement, empowerment, and active participation in the decision making process.

This is a clinical multicenter, non-randomized, interventional phase II study involving Danish surgical departments planned to commence in the first quarter of 2024. The aim of the study is to examine whether shared decision making and using a patient decision aid (PtDA) in consultations affects patients' choice of management compared with historical data. The secondary aim is to investigate Patient Reported Experience Measures (PREMs) and Patient Reported Outcome Measures (PROMs) using questionnaire feedback directly from the patients.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically verified malignant colorectal polyp removed endoscopically and CT-scan (and MRI if the malignant polyp was situated in the rectum) shows N0, M0 disease.

Exclusion Criteria:

* Inability to provide informed consent
* Inoperable due to comorbidity
* Known residual tumor left in situ after local resection, >N0 or >M0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients undergoing completion surgery of an unexpected malignant polyp compared to historical data. | 30 days

SECONDARY OUTCOMES:
Rate of patients with an unexpected malignant polyp undergoing completion surgery without residual tumor or lymph node metastases compared to historical data. | 45 days
Number of patients with postoperative morbidity 30 days after surgery | 30 days postoperatively
Number of patients with postoperative mortality 30 days after surgery | 30 days postoperatively
Number of patients with postoperative morbidity 90 days after surgery | 90 days postoperatively
Number of patients with postoperative mortality 90 days after surgery | 90 days postoperatively
Number of patients with recurrence 3 years after cancer diagnosis | 3 years
Overall survival 3 years after cancer diagnosis | 3 years
Quality of life as measured by the the European Organization for Research and Treatment of Cancer Quality of Life questionnaire. | 24 hours after clinical encounter
  Score range 1-100. The higher the score, the better the quality of life.
Quality of life as measured by the European Organization for Research and Treatment of Cancer Quality of Life questionnaire. | 3 months after clinical encounter
  Score range 1-100. The higher the score, the better the quality of life.
Quality of life as measured by the European Organization for Research and Treatment of Cancer Quality of Life questionnaire. | 6 months after clinical encounter
  Score range 1-100. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Würtz, MD, Principal Investigator — Vejle Hospital, Center for Shared Decision Making and Surgical Department; Karina D Steffensen, Prof PhD MD, Study Chair — Center For Shared Decision Making, Vejle Hospital; Hans B Rahr, Prof Dr MD, Study Chair — Surgical Department, Vejle Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wurtz HJ, Rahr HB, Lindebjerg J, Edwards A, Steffensen KD. Impact of an in-consult patient decision aid on treatment choices and outcomes of management for patients with an endoscopically resected malignant colorectal polyp: a study protocol for a non-randomised clinical phase II study. BMJ Open. 2023 Nov 14;13(11):e073900. doi: 10.1136/bmjopen-2023-073900. PMID 37963688